CLINICAL TRIAL: NCT01350375
Title: A Randomized Double-Blind Placebo Controlled Multi-Center Study to Evaluate the Safety and Efficacy of Botulinum Neurotoxin Type A in the Treatment of Forward Head Posture With Associated Episodic Headache Disorder
Brief Title: Safety and Efficacy Study of Botox in the Treatment of Forward Head Posture With Associated Episodic Headache Disorder
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: The Research Center of Southern California (Other)
Responsible Party: Principal Investigator, April Tenorio, Principal Investigator, The Research Center of Southern California
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: BTX0805
Record Dates: First submitted 2011-05-06; First posted 2011-05-09 (Estimated); Last update posted 2019-09-11 (Actual); Status verified 2019-09

CONDITIONS: Forward Head Posture With Associated Episodic Headache Disorder
MeSH Terms: interventions — Botulinum Toxins, Type A; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Saline (Placebo Comparator)
  Interventions: Drug: Saline
- Botox (Active Comparator)
  Interventions: Drug: Botox

INTERVENTIONS:
Drug: Botox
  Arms: Botox
Drug: Saline
  Arms: Saline

SUMMARY:
This study will investigate the therapeutic utility of BOTOX in reducing the degree of Forward Head Posture (FHP) with associated headache and myofascial pain, decreasing the frequency of headache, and improving the overall quality of life.

DETAILED DESCRIPTION:
This is a multi-center, prospective, double-blind, placebo-controlled parallel study investigating the use of BOTOX in the treatment of patients with FHP and associated headache using a novel fixed site injection paradigm.

Fifteen subjects will be randomized to receive BOTOX® and fifteen will receive placebo injections. Study subjects will receive one cycle of injections, up to a maximal total dosage of 250U. The study duration is approximately 4 months and is composed of a Screening Visit (Visit 1, Month -1), a Baseline Visit (Visit 2, Day 0), and three Follow-Up Visits 1 month apart (Months 1, 2 and 3).

ELIGIBILITY:
Inclusion Criteria:

1. Outpatient, healthy male or female volunteers of any race, >18 years of age. Females of childbearing potential must have a negative urine pregnancy test result at the Baseline Visit and practice a reliable method of contraception throughout the study;

   A female is considered of childbearing potential unless she is:
   * postmenopausal for at least 12 months prior to study drug administration;
   * without a uterus and/or both ovaries; or
   * has been surgically sterile for at least 6 months prior to study drug administration.

   Reliable methods of contraception are:
   * hormonal methods must be started at least 90 days prior to study drug administration
   * intrauterine device in use > 30 days prior to study drug administration; or
   * barrier methods plus spermicide in use at least 14 days prior to study drug administration.
   * partner has had a vasectomy at least 3 months previously or a confirmatory 0 sperm count test.

     * Female subjects of childbearing potential who are not sexually active are not required to practice a reliable method of contraception. They may be enrolled at the Investigator's discretion provided that they are counseled to remain sexually inactive for the duration of the study and understand the possible risks involved in getting pregnant during the study.
2. Diagnosis of FHP with at least two-fingerbreadth head forward posture.
3. Episodic Headache Disorder as per the following criteria:

   * < 15 headache days per month including 10-14 days/month episodic migraine (with or without aura);
   * Chronic migraine is excluded;
   * Chronic Tension type HA is excluded.
4. Subjects able to understand the requirements and participate in the study, including completing questionnaires, maintaining a Headache Diary, signing Informed Consent, and authorizing the use/release of health and research study information.

Exclusion Criteria:

1. Pregnant (positive urine pregnancy test), planning to become pregnant during the study period, breast-feeding, or of childbearing potential and not practicing reliable contraception.
2. Patients with clinically significant spinal abnormalities (e.g., scoliosis).
3. Presence of cervical dystonia.
4. Medical condition that may increase risk of exposure to botulinum toxin (e.g., Myasthenia Gravis, Eaton-Lambert Syndrome, Amyotrophic Lateral Sclerosis, or any other disease that might interfere with neuromuscular function).
5. Use of aminoglycoside antibiotics, curare-like agents, or other agents that might interfere with neuromuscular function.
6. Injection Site Issues: profound atrophy or excessive muscle weakness in the target areas of injection, skin problems or infection at any of the injection sites.
7. Subjects with an allergy or sensitivity to any component of BOTOX® (Section 5.2).
8. Evidence of recent alcohol/drug abuse.
9. History of poor cooperation, non-compliance with medical treatment, or unreliability.
10. Uncontrolled systemic disease, condition or situation that, in the investigator's opinion, may put the subject at significant risk, confound study results, or significantly interfere with study participation, and/or life expectancy less than 12 months
11. Participation in an investigational drug or device study within 30 days of the Screening/Baseline Visit.
12. Administration of BOTOX® within the last 3 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2009-09; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Determining the efficacy and safety of BOTOX injections • The change in number of headache free days; • % days with headache; • Average headache severity; • Number of headache episodes (number of headaches). | 4 months
  The primary objective of this study is to determine the efficacy and safety of BOTOX injections in the treatment of forward head posture with associated Episodic Headache Disorder through:
  * The change in number of headache free days;
  * % days with headache;
  * Average headache severity;
  * Number of headache episodes (number of headaches).

SECONDARY OUTCOMES:
Determining the efficacy and safety of BOTOX injections | 4 months
  * To determine the efficacy and safety of BOTOX injections on the change in forward head posture as measured by the improvement in the degree of FHP (measured in cm and finger breadths) at the primary analysis point of 8 weeks post-injection.
  * To determine the efficacy and safety of BOTOX injections on the change in myofascial pain measured on visual analog scale scores.

CONTACTS AND LOCATIONS:
Locations (1):
- The Research Center of Southern California, Oceanside, California, United States